CLINICAL TRIAL: NCT01006629
Title: A Prospective, Multicenter, Open-label, Non-comparative Study of Safety and Efficacy of Synagis in Children at High Risk of Severe Respiratory Syncytial Virus Infection in the Russian Federation
Brief Title: Palivizumab for Prevention of Severe Respiratory Syncytial Virus Infection in Russian Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Konstantin Gudkov, Clinical Research Project Manager, Abbott Laboratories LLC Russia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: W10-664
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-06

CONDITIONS: Respiratory Syncytial Virus Infection; Premature Birth; Bronchopulmonary Dysplasia; Congenital Heart Disease
Keywords: Efficacy of palivizumab; Respiratory syncytial virus (RSV) infection; Prevention of severe RSV infection; Preterm infants; Infants with bronchopulmonary dysplasia; Infants with hemodynamically significant congenital heart disease
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Premature Birth; Bronchopulmonary Dysplasia; Heart Defects, Congenital; Infections | interventions — Palivizumab

ARMS (1):
- palivizumab (Experimental): palivizumab 15 mg/kg intramuscularly every 30 days for 3 to 5 injections
  Interventions: Biological: palivizumab

INTERVENTIONS:
Biological: palivizumab — palivizumab 15 mg/kg intramuscularly
  Other Names: ABT-315 (MEDI-493); Synagis 15 mg/kg intramuscularly

SUMMARY:
100 Russian children of 2 years of age and less in high-risk populations (preterm, and/or with heart and lung problems) will receive palivizumab (Synagis) 15 mg/kg intramuscularly as prophylaxis to severe respiratory syncytial virus (RSV) infection in order to study the safety and efficacy of the drug in Russian subjects.

DETAILED DESCRIPTION:
A prospective, multicenter, open-label, non-comparative study of safety and efficacy of palivizumab (Synagis) 15 mg/kg intramuscularly as prophylaxis to severe lower respiratory tract respiratory syncytial virus infection in 100 Russian children of 2 years of age and less in high-risk populations (preterm infants [less than or equal to 35 weeks gestational age], infants with bronchopulmonary dysplasia [BPD], and infants with hemodynamically significant congenital heart disease [HSCHD]).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled into the study:

1. Infants at high risk of severe RSV infection defined as fulfilling at least one of the following:

   * Infants born at less than or equal to 35 weeks gestational age AND are less than or equal to 6 months of age at enrollment
   * Infants less than or equal to 24 months of age at enrollment AND with a diagnosis of bronchopulmonary dysplasia (defined as oxygen requirement at a corrected gestational age of 36 weeks) requiring intervention/management (i.e., oxygen, diuretics, bronchodilators, corticosteroids, etc.) anytime within 6 months prior to enrollment
   * Infants less than or equal to 24 months of age at enrollment with hemodynamically significant congenital heart disease, either cyanotic or acyanotic, unoperated or partially corrected. Children with acyanotic cardiac lesions must have pulmonary hypertension (greater than or equal to 40 mmHg measured pressure in the pulmonary artery [ultrasound acceptable]) or the need for daily medication to manage congenital heart disease. Children with the following conditions are not eligible: hemodynamically insignificant small atrial or ventricular septal defects, patent ductus arteriosis, children with aortic stenosis, pulmonic stenosis, or coarctation of the aorta alone.
2. Informed Consent Form signed by parent(s).

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for the study:

1. Hospitalization at the time of enrollment (unless discharge is anticipated within 14 days).
2. Mechanical ventilation (including continuous positive airway pressure [CPAP]) at the time of enrollment.
3. Life expectancy less than 6 months.
4. Active respiratory illness, or other acute infection.
5. Known renal impairment, as determined by the investigator.
6. Known hepatic impairment, as determined by the investigator.
7. History of seizures (except neonatal seizures).
8. Unstable neurological disorder (includes, but is not restricted to, epilepsy and decompensated hydrocephaly).
9. Known immunodeficiency, as determined by the investigator.
10. Allergy to immunoglobulin products.
11. Prior receipt of RSV vaccine or prophylaxis (e.g., palivizumab or motavizumab), or administration of a product possibly containing RSV-neutralizing antibody within 100 days prior to enrollment (includes, but is not restricted to, the following: RSV hyperimmunoglobulin, polyclonal intravenous immunoglobulin, cytomegalovirus hyperimmunoglobulin, varicella zoster hyperimmunoglobulin).
12. Participation in another clinical trial within 30 days prior to enrollment.
13. Previous enrollment in this trial.
14. For any reason, subject is considered by the investigator to be an unsuitable candidate for this study.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin M Gudkov, MD, Study Director — Abbott
Locations (19):
- Russia (19):
  - Site Ref # / Investigator 22699, Ivanovo
  - Site Ref # / Investigator 22694, Kazan'
  - Site Ref # / Investigator 24022, Moscow
  - Site Ref # / Investigator 15744, Moscow
  - Site Ref # / Investigator 15745, Moscow
  - Site Ref # / Investigator 24025, Moscow
  - Site Ref # / Investigator 15781, Moscow
  - Site Ref # / Investigator 22686, Moscow
  - Site Ref # / Investigator 15747, Moscow
  - Site Ref # / Investigator 22696, Novosibirsk
  - Site Ref # / Investigator 24023, Novosibirsk
  - Site Ref # / Investigator 22692, Saint Petersburg
  - Site Ref # / Investigator 22683, Saint Petersburg
  - Site Ref # / Investigator 22693, Saint Petersburg
  - Site Ref # / Investigator 22685, Saint Petersburg
  - Site Ref # / Investigator 15722, Saint Petersburg
  - Site Ref # / Investigator 15748, Saint Petersburg
  - Site Ref # / Investigator 15782, Saint Petersburg
  - Site Ref # / Investigator 15746, Tomsk

REFERENCES:
- [Derived] Turti TV, Baibarina EN, Degtiareva EA, Keshishyan ES, Lobzin YV, Namazova-capital VE, Cyrillicaranova LS, Prodeus AP, Gudkov KM, Kruglova AI, Schulz GA, Notario GF. A prospective, open-label, non-comparative study of palivizumab prophylaxis in children at high risk of serious respiratory syncytial virus disease in the Russian Federation. BMC Res Notes. 2012 Sep 4;5:484. doi: 10.1186/1756-0500-5-484. PMID 22943074
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=23151&CFID

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled into the study in 3 geographic areas of the Russian Federation. Recruitment began in November 2009 and ended in December 2009. Subjects at high risk of severe RSV infection (including preterm infants, infants with BPD, and infants with HSCHD) were identified as candidates for the study on the basis of routine assessments.
Period: Overall Study
Arm/Group | Palivizumab
Started | 100
Completed | 94
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Parent refused to continue participation | 1
Not completed — Parent unable to perform site visit | 4

BASELINE CHARACTERISTICS:
Arm/Group | Palivizumab
Number analyzed (Participants) | 100
Age Continuous [Mean (Standard Deviation); unit: months] | 8.2 (6.3)
Age, Customized [Number; unit: participants]
  Between 0 and 3 months | 28
  Between 4 and 6 months | 24
  Between 7 and 9 months | 14
  Between 10 and 12 months | 7
  Between 13 and 15 months | 8
  Between 16 and 18 months | 10
  Between 19 and 21 months | 5
  Between 22 and 24 months | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 48
Region of Enrollment [Number; unit: participants]
  Russian Federation | 100
Gestational Age [Mean (Standard Deviation); unit: weeks] — Gestational age is defined as the time from mother's last menstrual period until birth.
  weeks | 33.4 (5.1)
Gestational Age, categorical [Number; unit: participants]
  Less than 29 weeks gestational age | 23
  Between 29 and 32 weeks gestational age | 22
  Between 33 and 35 weeks gestational age | 22
  Greater than 35 weeks gestational age | 33
Infants born <= 35 weeks gestational age and <= 6 months of age at enrollment [Number; unit: participants]
  Yes | 33
  No | 67
Infants <= 24 months of age at enrollment and with a diagnosis of BPD [Number; unit: participants]
  Yes | 46
  No | 54
Infants <= 24 months of age at enrollment and with HSCHD [Number; unit: participants]
  Yes | 30
  No | 70

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: Treatment-emergent adverse events were defined as those occurring after study drug initiation and within 30 and 100 days after the last dose of study drug. The number of subjects experiencing a serious or nonserious treatment-emergent adverse event within 30 days after the last dose of study drug is summarized. See the Reported Adverse Events section for details.
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 100
participants | 41

2. Primary Outcome: Number of Hospitalizations Due to Respiratory Syncytial Virus (RSV)
Description: Number of subjects experiencing an RSV hospitalization
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 100
participants | 0 [0.0 to 3.6]

3. Secondary Outcome: Total Number of RSV Hospitalization Days
Description: All secondary outcome measures were related to hospitalization due to RSV infection. No RSV hospitalizations occurred during the study; therefore, evaluation of the secondary outcome measures was not possible.
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Total RSV Hospitalization Days With Increased Supplemental Oxygen Requirement
Description: as for outcome 3
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Intensive Care Unit (ICU) Admissions During RSV Hospitalization
Description: Outcome measure refers to the number of subjects admitted to the ICU during RSV hospitalization. No RSV hospitalizations occurred during the study; therefore, evaluation of the secondary outcome measures was not possible.
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Total Days of RSV ICU Stay
Description: as for outcome 3
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Subjects Who Received Mechanical Ventilation During RSV Hospitalization
Description: as for outcome 3
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Total Days of Mechanical Ventilation During RSV Hospitalization
Description: as for outcome 3
Time Frame: Through 30 days following the last injection of palivizumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug through 100 days after the last dose of study drug
Arm/Group | Palivizumab
Serious Adverse Events (participants affected / at risk) | 10/100
Other Adverse Events (participants affected / at risk) | 39/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=100)
Supraventricular tachycardia (Cardiac disorders) | 1
Enteritis (Gastrointestinal disorders) | 3
Bronchitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=100)
Arrhythmia (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Anal stenosis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Food allergy (Immune system disorders) | 1
Ascariasis (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Dacryocystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 19
Upper respiratory tract infection (Infections and infestations) | 8
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Nervousness (Psychiatric disorders) | 2
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study had no control group; relative comparisons are only possible with current product information for palivizumab. No RSV hospitalizations occurred during the study; therefore, secondary outcome measures could not be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.